CLINICAL TRIAL: NCT02081040
Title: Cross Sectional Observation Study of Cough Dysfunction in Infratentorial Brain Lesion Patients, as Assessed by M-mode Sonography
Brief Title: Coughing in Infratentorial Brain Lesion Patients
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sun Im, Assistant Professor, The Catholic University of Korea
Other Study IDs: HC 13OISE0066_1
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Stroke
Keywords: brainstem; diaphragm; deglutition disorder; sonography
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Infratentorial dysphagia patients: Infratentorial brain lesion patients with confirmed evidence of dysphagia
- Supratentorial dysphagia patients: Supratentorial brain lesions\ patients with confirmed evidence of dysphagia
- Brain lesion patients without dysphagia: Brain lesion patients with no evidence of dysphagia
  Interventions: Other: Not applicable (observational study with no active intervention)

INTERVENTIONS:
Other: Not applicable (observational study with no active intervention)
  Groups: Brain lesion patients without dysphagia

SUMMARY:
To record diaphragm excursion in infratentorial brain lesions patients with dysphagia during coughing and compare them to those with supratentorial brain lesion patients with dysphasia and those with no dysphagia at a university affiliated rehabilitation department.

DETAILED DESCRIPTION:
Our previous work has shown that stroke patients with dysphagia have impaired diaphragm excursion in comparison to those with no dysphagia. It has been postulated that respiratory and cough function are primarily controlled by respiratory and swallowing centers located in the brainstem.We postulated that those with infratentorial brain lesions would have more impaired cough and respiratory function than those with non-brainstem lesions and supratentorial brain lesions.

However there has been no studies whether those with infratentorial brain lesions have more impaired cough function and decreased diaphragm excursion than those with supratentorial brain lesions.

ELIGIBILITY:
Inclusion Criteria:

Group 1- Brainstem lesion subjects with dysphagia that would require insertion of a nasogastric tube Group 2- Non-brainstem lesion subjects with dysphagia that would require insertion of a nasogastric tube Group 3- Stroke patients with no evidence of dysphagia

Exclusion Criteria:

* Episode of acute pneumonia or pulmonary embolism at time of enrollment
* Previous history of chronic respiratory disorders or other systemic disorders that may affect respiratory function ( ex, rheumatoid arthritis, chronic renal disease, spinal cord injury)
* Stroke patients with multiple brain lesions
* Episode of Diaphragm weakness due to peripheral polyneuropathy or unilateral phrenic nerve palsy
* Previous episode of abdominal or thoracic surgery within one year of enrollment
* Concomitant diagnosis of myopathy, muscular dystrophy or other disorders that may affect respiratory muscles.
* Episode of rib fracture within one year of enrollment
* Chronic alcoholism
* Patient with previous diagnosis of dementia or with impaired cognitive function that may limit full participation at the evaluation
* Patient with tracheostomy state

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dysphagia patients due to brain lesions at a university affiliated hospital
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Diaphragm excursion | baseline one time
  Diaphragm excursion as assessed by m mode sonography

SECONDARY OUTCOMES:
Maximal inspiratory pressure | baseline one time
Peak cough flow force during voluntary coughing | baseline one time

OTHER OUTCOMES:
maximal expiratory pressure | baseline one time
spirometry findings | baseline one time
Cough force during reflexive coughing | baseline one time
  Peak flow force during reflexive coughing

CONTACTS AND LOCATIONS:
Overall Officials: Sun Im, MD PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Bucheon St Mary's Hospital, Bucheon-si, Gyonngido, South Korea